CLINICAL TRIAL: NCT04440761
Title: Barts Myocardial Infarction With Non-Obstructed Coronary Arteries (MINOCA) Registry
Brief Title: Barts-MINOCA Registry
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: REDA: 130386
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Infarction; Gender; Coronary Microvascular Disease
MeSH Terms: conditions — Myocardial Infarction; Coitus; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Troponin rise/ diagnosis of MINOCA: This study aims to assess, in a real-world setting, the safety, efficacy and feasibility of further investigations in patients diagnosed with MINOCA among all patients with coronary artery disease.
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — Observation only

SUMMARY:
The last 15 years the introduction of primary angioplasty has radically improved outcomes for acute myocardial infarction (AMI). However, the system wide availability of prompt investigation has revealed an important group of patients where progress has stalled, the diagnosis is unclear and therapeutic approaches are uncertain. Myocardial infarction with non-obstructive coronary arteries (MINOCA) is found in 1 - 13% of all patients with a clinical diagnosis of AMI.

These patients present a therapeutic predicament since coronary revascularization is not appropriate. Guidelines do not exist for their management - yet the condition is not benign - the 12-month prognosis, although better than obstructive coronary artery disease patients is still guarded with recent data suggesting many questions remain unanswered.

DETAILED DESCRIPTION:
This study utilises a prospectively collected clinical database. All patients referred to the Interventional Cardiology team are included onto this database. No patients will be contacted solely for research purposes. Patients will not have any investigations/procedures performed for research purposes. All data will only be available for access by named members of the Interventional Cardiology team. Data will be anonymised by the clinical care team and passed onto the research team before it is used and no patient identifiable information will be used in the analysis of the study or the publications of its results.

The database started in April 2015 and has collected data on all patients so far and will continue to do so for the duration of clinical work by the Interventional Cardiology team. As a result this study will continue indefinitely.

This study will include all patients admitted to or reviewed in clinic at Barts Health NHS Trust with either a diagnosis of MINOCA or who do not have a clear cause of a troponin rise. These patients range from young adults to the elderly and will include any patient ≥16 years of age. Patients who are followed up with and without any intervention (i.e. both medically managed patients as well as patients undergoing intervention) are equally as important and therefore the investigators shall include both groups of patients.

Patients will be included from referrals made by other clinicians either as in or outpatients. All these patients have their clinical data captured on a database or hospital based clinical programme.

This study aims to assess, in a real-world setting, the safety, efficacy and feasibility of further investigations in patients diagnosed with MINOCA among all patients with coronary artery disease.

The study will test various hypothesis including but not limited to:

1. The efficacy of diagnosis rates of CMR in patients diagnosed with MINOCA
2. Outcomes in patients diagnosed with MINOCA treated medically
3. Long-term outcome of patients diagnosed with MINOCA

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients ≥16 years of age will be included
* All patients will have a diagnosis MINOCA. Any patient who does not have a clear cause of troponin rise

Exclusion Criteria:

* Patients <16 years will not be included in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients admitted to or reviewed in clinic at Barts Health NHS Trust with either a diagnosis of MINOCA or who do not have a clear cause of a troponin rise. These patients range from young adults to the elderly and will include any patient ≥16 years of age. Patients who are followed up with and without any intervention (i.e. both medically managed patients as well as patients undergoing intervention) are equally as important and therefore we shall include both groups of patients.
  Patients will be included from referrals made by other clinicians either as in or outpatients. All these patients have their clinical data captured on a database or hospital based clinical programme.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Assessment of mortality
Mortality | 1 year
  Assessment of mortality
Formal diagnosis made of the cause of troponin rise | Baseline
  Diagnosis
Timing of diagnosis made of the cause of troponin rise | Baseline
  Time to first diagnosis
Questionnaire to assess change in symptoms at 2 months post-initial review in clinic/ward | 2 months
  Change in symptoms assessed by Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jones, MBBS, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No